CLINICAL TRIAL: NCT07253935
Title: Efficacy of a Combined Approach of Therapeutic Exercise, Psychotherapy, and Therapeutic Education in Patients With Depression: The ACTIDEP Randomized Controlled Trial
Brief Title: Impact of Therapeutic Exercise Integrated With Psychotherapy and Education in Patients With Depression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MarcoMateoRiera (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACTIDEP2025RCT
Record Dates: First submitted 2025-11-18; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Depression Disorder
Keywords: Mental disorders; Depression; Exercise; Physical activity
MeSH Terms: conditions — Mental Disorders; Depression; Motor Activity | interventions — Psychotherapy; Acceptance and Commitment Therapy; Cognitive Behavioral Therapy; Exercise; Educational Status; Exercise Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants and care providers cannot be masked due to the nature of the exercise intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychotherapy (Active Comparator): Conventional psychotherapy for the treatment of depression.
  Interventions: Behavioral: Psychotherapy
- Exercise, therapeutic education and psychotherapy (Experimental): Graded activity in combination with exercise, therapeutic education and psychotherapy
  Interventions: Behavioral: Psychotherapy; Behavioral: Graded activity combined with exercise and education

INTERVENTIONS:
Behavioral: Psychotherapy — Conventional psychotherapy for depression, including Acceptance and Commitment Therapy, Behavioral Activation, Cognitive Behavioral Therapy, Interpersonal Therapy, and Mindfulness-Based Cognitive Therapy.
  Other Names: Acceptance and Commitment Therapy; Behavioral Activation; Cognitive Behavioral Therapy
Behavioral: Graded activity combined with exercise and education — This intervention consists of a graded activity program combined with exercise and therapeutic education in motor behavior to improve physical activity levels, self-efficacy and mood
  Other Names: Biobehavioral physiotherapy; Therapeutic education; Exercise Therapy
  Arms: Exercise, therapeutic education and psychotherapy

SUMMARY:
The goal of this clinical trial is to evaluate whether a combined approach including therapeutic exercise, psychotherapy, and therapeutic education can improve depressive symptoms and quality of life in adults diagnosed with depression.

The main questions it aims to answer are:

Does a biobehavioral intervention that integrates exercise, psychotherapy, and education reduce depressive symptoms more effectively than psychotherapy alone? Does this combined approach improve quality of life, physical function, and sleep quality compared with standard psychological therapy? Researchers will compare the intervention group (therapeutic exercise + psychotherapy + education) to the control group (psychotherapy alone) to determine whether the integrated program provides greater improvements in mental health and well-being.

Participants will:

Complete an initial assessment including demographic data, physical tests, and validated questionnaires.

Be randomly assigned to one of the two groups. If in the intervention group, take part in an 8-week telematic program consisting of graded activity, therapeutic exercise, and educational sessions.

Undergo post-intervention assessments and a follow-up evaluation 12 weeks after the program ends.

This study aims to provide evidence on whether combining therapeutic exercise and education with psychotherapy can enhance treatment outcomes and promote long-term adherence to physical activity in people with depression.

DETAILED DESCRIPTION:
Depressive disorder is one of the most prevalent and disabling mental health conditions worldwide. Although pharmacological and psychological treatments remain the cornerstone of care, many patients continue to experience residual symptoms, recurrent episodes, or limitations in daily functioning and quality of life. In recent years, exercise-based interventions have gained recognition as a valuable adjunct to conventional treatment, showing beneficial effects on mood regulation, physical health, and overall well-being. Nonetheless, the most effective ways to integrate structured exercise, therapeutic education, and psychotherapy within a coordinated, patient-centered framework are still not well established.

This randomized controlled trial aims to examine the effects of a biobehavioral physiotherapy program that combines graded activity, therapeutic exercise, and patient education delivered concurrently with conventional psychotherapy. The rationale for this combined approach lies in addressing both physical and behavioral components of depression through a structured, progressive, and individualized program. Graded activity is designed to progressively increase patient´s tolerance to physical effort and promote engagement in meaningful daily tasks, while therapeutic education targets maladaptive beliefs about pain, fatigue, and activity avoidance. Together, these components aim to enhance self-efficacy, functional performance, and adherence to recovery-oriented behaviors.

The intervention will be delivered online under professional supervision, ensuring accessibility and continuity of care. The program will last eight weeks and will include structured exercise sessions emphasizing strength, mobility, and aerobic capacity, as well as educational modules focused on pacing, goal setting, and self-management strategies. The use of telehealth enables real-time monitoring, feedback, and personalized adjustments to exercise dosage and progression. Participants in the control group will continue receiving conventional psychotherapy for depression, following their regular clinical routine.

To ensure methodological rigor, randomization will be computer-generated with a 1:1 allocation ratio. Outcome assessments will be conducted by an independent evaluator blinded to group allocation. Standardized and validated measures will be used to assess depressive symptoms, quality of life, physical activity levels, functional capacity, self-efficacy, and sleep quality. Assessments will occur at baseline, mid-intervention, post-intervention, and 12-week follow-up to capture both immediate and sustained effects of the program.

Data will be analyzed following an intention-to-treat approach. Analysis of covariance (ANCOVA) and repeated-measures models will be applied to determine between-group differences and time-by-group interactions, adjusting for baseline scores and potential covariates. Effect sizes will be calculated to estimate the magnitude of the observed effects.

This study is expected to contribute to the growing body of evidence supporting integrative, biobehavioral approaches to the management of depression. By combining exercise and education within a psychotherapeutic framework, the program seeks to promote behavioral activation, enhance perceived control, and improve overall quality of life. If effective, this model could serve as a scalable, cost-effective, and accessible intervention for patients with depressive disorders, expanding the role of physiotherapy and interdisciplinary collaboration in mental health care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of depression or dysthymia according to the ICD-11 criteria (including unspecified depressive disorder, code 6A7Z) or DSM-5-TR criteria confirmed by their referring physician.
* A patient currently undergoing psychological treatment for depression with a score above the established cutoff in a validated depression questionnaire.

Exclusion Criteria:

* Pregnancy.
* Presence of neurological comorbidities or neurological signs.
* Systemic rheumatic diseases, including fibromyalgia.
* Central nervous system disorders.
* Severe cognitive impairment.
* Schizophrenia, psychotic disorders, or bipolar spectrum disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms | From enrollment to the end of treatment at 8 weeks, with follow-up 12 weeks after completion of treatment.
  The Patient Health Questionnaire-9 (PHQ-9) will be used to assess depressive symptoms. This is a self-administered questionnaire with nine items scored on a four-point Likert scale (0-3). Higher scores indicate greater severity.
Quality of life | From enrollment to the end of treatment at 8 weeks, with follow-up 12 weeks after completion of treatment.
  The World Health Organization Quality of Life Questionnaire (WHOQoL-BREF) is a self-administered instrument validated in Spanish that assesses perceived quality of life across different domains. It consists of 26 items rated on a 5-point Likert scale, yielding a total score and four domain scores: physical health, psychological health, social relationships, and environment. Scores are transformed to a 0-100 scale, with higher scores indicating better quality of life

SECONDARY OUTCOMES:
Physical activity levels | From enrollment to the end of treatment at 8 weeks, with follow-up 12 weeks after completion of treatment.
  The Global Physical Activity Questionnaire (GPAQ) is a self-administered instrument that assesses physical activity across three domains: work-related activity, transportation, and recreational activity. It consists of 16 items that estimate the time spent in different intensities of activity (light, moderate, and vigorous), with results expressed in MET-minutes per week
Sleep quality | From enrollment to the end of treatment at 8 weeks, with follow-up 12 weeks after completion of treatment
  The Pittsburgh Sleep Quality Index (PSQI) is a valid and reliable instrument (α = 0.76) used to assess sleep quality. It consists of 19 self-reported items evaluating seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each component is scored from 0 to 3, yielding a total score ranging from 0 to 21, with higher scores indicating poorer sleep quality. A global score greater than 5 suggests clinically relevant sleep disturbances.
Lower limb strength | From enrollment to the end of treatment at 8 weeks, with follow-up 12 weeks after completion of treatment
  The 30-Second Chair-Stand Test (30s-CST) is a validated functional test designed to assess lower-limb muscle strength and endurance. It consists of counting the number of times an individual can rise fully from a standard chair without using their arms within a 30-second period. A standard chair (43-45 cm high) is used, with the participant seated upright, feet flat on the floor and arms crossed over the chest.
  The outcome is expressed as the total number of correctly completed repetitions within 30 seconds, with higher scores indicating greater lower-limb strength and endurance.
Maximal oxygen uptake (V̇O2Max) | From enrollment to the end of treatment at 8 weeks, with follow-up 12 weeks after completion of treatment
  The Chester Step Test (CST) is a progressive submaximal test used to estimate maximal oxygen uptake (V̇O2Max). It involves stepping up and down on a fixed-height bench (typically 25-30 cm for most adults) following a progressively increasing pace set by a metronome or audio recording.
  The test consists of five two-minute stages, with cadence increasing at each stage until the participant reaches 80% of their age-predicted maximum heart rate (220-age) or is unable to maintain the required pace. Throughout the test, heart rate and ratings of perceived exertion (RPE, Borg 6-20 scale) are recorded at the end of each stage.With this information VO2Max values are estimated.
  Unit of measure: mlO2/kg/min
Self-Efficacy to Regulate Exercise | From enrollment to the end of treatment at 8 weeks, with follow-up 12 weeks after completion of treatment
  The Self-Efficacy Questionnaire to Regulate Exercise (SEQRE) is a valid and reliable instrument (α = 0.84) consisting of 7 items that assess participants' confidence in maintaining a regular exercise routine (three or more times per week). Each item is rated on a scale from 0 ("I cannot do it at all") to 100 ("I am very confident I can do it"), with higher scores indicating greater perceived self-efficacy for exercise practice

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Diez-Quevedo C, Rangil T, Sanchez-Planell L, Kroenke K, Spitzer RL. Validation and utility of the patient health questionnaire in diagnosing mental disorders in 1003 general hospital Spanish inpatients. Psychosom Med. 2001 Jul-Aug;63(4):679-86. doi: 10.1097/00006842-200107000-00021. PMID 11485122
- [Background] Favela Ramírez, C. A., Castro Robles, A. I., Bojórquez Díaz, C. I., & Chan Barocio, N. L. (2022). Propiedades psicométricas del índice de calidad de sueño de Pittsburgh en deportistas. riccafd: Revista Iberoamericana de Ciencias de la Actividad Física y el Deporte, 11(3), 29-46. https://dialnet.unirioja.es/servlet/articulo?codigo=8736227
- [Background] Lein DH Jr, Alotaibi M, Almutairi M, Singh H. Normative Reference Values and Validity for the 30-Second Chair-Stand Test in Healthy Young Adults. Int J Sports Phys Ther. 2022 Aug 1;17(5):907-914. doi: 10.26603/001c.36432. eCollection 2022. PMID 35949374